CLINICAL TRIAL: NCT05616052
Title: Prospective Randomized Controlled Study on the Improvement of Body Weight Among Overweight and Obese Patients Through Different Smeglutide Administration Methods
Brief Title: Comparison of Body Weight Change Through Different Smeglutide Administration Methods
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, xiaolong zhao, Professor of endocrinology department, Shanghai Public Health Clinical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-10-weight loss-SPHCC
Record Dates: First submitted 2022-10-05; First posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Weight Change, Body
MeSH Terms: conditions — Body Weight Changes | interventions — semaglutide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard arm (Active Comparator): standard arm will start from 0.25mg per week for four weeks, then increase to 0.5mg per week for four weeks, and 1mg per week maintenance dose for 8 weeks..
  Interventions: Drug: Semaglutide
- titration arm (Active Comparator): Titration arm dosage regime depends on the tolerance of the semaglutide from patients. The dosage will stabilize on the dose which patients could tolerate
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — treatment with different dosage regimes
  Other Names: dosage regime

SUMMARY:
Investigators determined to detect the effect of smeglutide on body weight and metabolic indexes among overweight and obese participants through two different dosing programs.

DETAILED DESCRIPTION:
Participants will be randomized into either group. One group will start from 0.25mg per week for four weeks, then increase to 0.5mg per week for four weeks, and 1mg per week maintenance dose for 8 weeks. The other group dosage regime depends on the tolerance of the semaglutide from participants. The dosage will stabilize on the dose how much participant could tolerate. At the end of 16 weeks treatment, comparison will be carried out on weight change before and after treatment and (1) Comparison of different administration methods (standards and titrations) on participant compliance, appetite and quality of life improvement; (2) Comparison of metabolism (waist hip circumference, body fat and body composition, blood pressure, blood lipid, blood glucose, insulin resistance) in different administration modes; (3) Comparison of adverse reactions of metabolic drugs in different administration modes.

ELIGIBILITY:
Inclusion Criteria:

1. 18 ≤ age<75;
2. Overweight or obesity: meet either one of the following standards

   1. Patients with BMI ≥ 24 kg/m2 and at least one obesity complication (hypertension, hyperlipidemia, apnea syndrome, cardiovascular disease)
   2. Simple obese patients with BMI ≥ 28kg/m2
   3. Abdominal obesity, waist circumference ≥ 90 cm for males and ≥ 80 cm for females

Exclusion Criteria:

1. Have a personal or family history of medullary thyroid carcinoma (MTC) or have multiple endocrine neoplasia type 2 (MEN-2) patients.
2. Patients with severe hypersensitivity to smeglutide or any other excipient component.
3. Diabetic patients (glycosylated hemoglobin ≥ 6.5% or fasting blood glucose ≥ 7.0 mmol/L or blood glucose ≥ 11.1 mmol/L 2 hours after meal or random blood glucose ≥ 11.1 mmol/L).
4. Triglyceride>5.6mmol/L;
5. Participants in other clinical drug trials in recent three months.
6. The range of weight change in recent 90 days is>5kg.
7. Cushing's syndrome and abnormal thyroid function.
8. Pregnant or breastfed women.
9. The study doctor judged that it was not suitable to participate in the test.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
weight change in kilograms | 16 weeks
  weight change in kilograms before and after treatment

SECONDARY OUTCOMES:
patient compliance in rate | 16 weeks
  rate of participants dropout of the study（in percentage)
waist hip circumference in centimeter | 16 weeks
  waist hip circumference in centimeter
number of adverse events | 16 weeks
  number of adverse events including hypoglycemia, nausea, vomiting, abdominal pain, diarrhea, constipation, indigestion, burping, flatulence, injection site allergy. Adverse reactions will recorded in percentage (number of participants developed particular adverse reaction divided by all participants in each group, % )
appetite change in score | 16 weeks
  appetite change measures in appetite questionnaire (visual analogue scales in assessment of appetite sensations, Units on scale is millimeter)
quality of life improvement in score | 16 weeks
  quality of life improvement (in WHOQOL~BREF, Units on scale is point);
body fat in percentage | 16 weeks
  body fat in percentage
body composition of lean mass in kilogram | 16 weeks
  body composition in kilogram of lean mass
blood pressure in mmHg | 16 weeks
  blood pressure in mmHg
blood lipid in concentration | 16 weeks
  blood lipid in including (total cholesterol, triglyceride, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol in mmol/L),
fasting blood glucose level | 16 weeks
  fasting blood glucose in milli-mole per liter
HOMA-Beta value | 16 weeks
  the value of 20 × FINS/（FBG-3.5）
total cholesterol in mmol/L | 16 weeks
  total cholesterolin mmol/L
triglyceride | 16 weeks
  triglyceride in mmol/L
low-density lipoprotein cholesterol | 16 weeks
  low-density lipoprotein cholesterol in mmol/L
high-density lipoprotein cholesterol | 16 weeks
  high-density lipoprotein cholesterol in mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: xiaolong zhao, Principal Investigator — Shanghai Public Health Clinical Center
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Y, Zhao L, Gao L, Pan A, Xue H. Health policy and public health implications of obesity in China. Lancet Diabetes Endocrinol. 2021 Jul;9(7):446-461. doi: 10.1016/S2213-8587(21)00118-2. Epub 2021 Jun 4. PMID 34097869
- [Background] Flint A, Raben A, Blundell JE, Astrup A. Reproducibility, power and validity of visual analogue scales in assessment of appetite sensations in single test meal studies. Int J Obes Relat Metab Disord. 2000 Jan;24(1):38-48. doi: 10.1038/sj.ijo.0801083. PMID 10702749
- [Background] Blundell J, Finlayson G, Axelsen M, Flint A, Gibbons C, Kvist T, Hjerpsted JB. Effects of once-weekly semaglutide on appetite, energy intake, control of eating, food preference and body weight in subjects with obesity. Diabetes Obes Metab. 2017 Sep;19(9):1242-1251. doi: 10.1111/dom.12932. Epub 2017 May 5. PMID 28266779